CLINICAL TRIAL: NCT05902273
Title: The Value of Peripheral Arterial Resistive Index in Evaluation of Tissue Perfusion in Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: Bezmialem V U
Record Dates: First submitted 2023-05-27; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Shock, Septic
Keywords: Septic shock; SBRI; SVRI; systemic vascular resistance index; resistive index; Pourcelot index
MeSH Terms: conditions — Shock, Septic | interventions — Hemodynamic Monitoring; Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- septic shock patients: mechanically ventilated septic shock patients
  Interventions: Diagnostic Test: hemodynamic monitoring; Diagnostic Test: resistive index; Diagnostic Test: Pleth variability index

INTERVENTIONS:
Diagnostic Test: hemodynamic monitoring — Baxter Starling Monitor for measuring cardiac output and systemic vascular resistance (SVRI) which is using bioreactance technology. We need to place four electrodes on chest wall (upper left, upper right, down left, down right) and input monitor demographic parameters. Also enter mean arterial pressure (MAP) for calculating SVRI so we input MAP every minute.Patient bed set as 45 degree head elevated and legs 0 degree. Just after start measuring, monitor needs to synchronize itself for patient. After synchronisation we start fluid challenge with passive leg raising option. This test has two stages. First stage calculating baseline parameters which takes 3 minutes and second stage is measuring difference with fluid challenge which also takes 3 minutes. At the end of first stage monitor shows to perform passive leg raise and we perform trendelenburg maneuver till head comes to 0 degree. After second stage measurement has finished.
  Other Names: Non Invasive Cardiac Output Monitor (NICOM)
Diagnostic Test: resistive index — We use ultrasonography at the same time with cardiac output monitor in both stages. First we determine the location of radial artery at wrist snuffbox at 1.5 centimeters depth with linear probe and confirm pulsatile flow with color mode. In Starling's baseline stage we measure and calculate resistive index with doppler P-mode in triplex setting 3 times. When received 3 same result successively we noted as SBRI-1. Second measurement is initiated at last 30 seconds of passive leg raising as described before and we noted our measurement as SBRI-2
  Other Names: SBRI; Snuffbox resistive index; Pourcelot index; doppler ultrasonography
Diagnostic Test: Pleth variability index — During all stages Masimo Rad-87 rainbow probe is placed patients index or middle finger and we note PVI-1 and PVI-2 at the same time with SBRI-1 and SBRI-2
  Other Names: PVI; Rad-87

SUMMARY:
In patients with septic shock, routine arterial blood pressure and central venous pressure are monitored in ICU. Conventional methods such as blood pressure and central venous pressure in septic patients cannot provide sufficient information in the follow-up due to the body's compensation mechanisms. The systemic vascular resistance index, which can be measured invasively or non-invasively with advanced hemodynamic monitoring methods, is a parameter that plays an important role in the management of septic patients.

Resistive index (Pourcelot Index) is an ultrasonic measurement method used to evaluate tissue perfusion and microcirculation. Since peripheral tissue perfusion is impaired in septic patients, the investigators think resistive index may be useful for management of sepsis. There are studies in the literature on the use of resistive index in the follow-up of patients.

The study will be about whether there is a correlation between the systemic vascular resistance index measured by cardiac output measurement, which is one of the advanced monitoring methods routinely used in the group requiring mechanical ventilation support in patients with septic shock, and the peripheral arterial resistive index, which is routinely used to evaluate tissue perfusion and microcirculation.

DETAILED DESCRIPTION:
Sepsis is not a specific disease but abnormal response for infection, leading to organ dysfunction. It is a clinical syndrome consisting of biological, biochemical, and physiological abnormalities which pathophysiology has not yet been fully determined. Sepsis is shaped by pathogenic factors and host factors (eg, gender, race and other genetic determinants, age, comorbidities, environment) and its features evolve over time. What distinguishes sepsis from infection is the presence of abnormal and/or irregular host response and organ dysfunction. It is one of the leading health problems worldwide and one of the leading causes of mortality in hospitalizations. Its estimated that there were 48.9 million cases and 11 million sepsis-related deaths worldwide in 2017, accounting for almost 20% of all global deaths. In an epidemiological study conducted in European intensive care units (ICU), the incidence of sepsis was reported as 38%. Pneumonia, urinary tract, and intra-abdominal infections account for more than 65% of all sepsis cases. According to the Surviving Sepsis Campaign (SSC) data, mortality rates in sepsis are 41% in Europe and 28.3% in the United States (USA). In a multicenter study involving 101,064 critically ill patients in Australia and New Zealand between 2002 and 2012, mortality rates due to sepsis were found to decrease over the years and finally to 18-20%. Recognition of sepsis, which can be very mortal, especially if not recognized fast and treatment not started, requires urgent attention.

Due to the lack of treatment options targeting microcirculatory and mitochondrial dysfunction, treatment has been focused on correcting the macrocirculatory dysfunction in addition to treating the underlying cause during septic shock. In the early phase of septic shock, external losses and hypovolemia are seen because of capillary leakage. Therefore, fluid resuscitation is often recommended to increase cardiac output and improve tissue perfusion. However, large boluses of fluids (>30 ml/kg) do not reliably increase blood pressure, urine output, and end-organ perfusion, and may lead to iatrogenic damage. Sepsis is characterized by disruptions in tissue perfusion and abnormal peripheral vascular resistance, because of disruptions in microcirculation. therefore, improving vascular function and organ damage is crucial in the management of septic shock. For treatment of hypotension; the need for fluid should be determined and the right amount of fluid resuscitation should be provided to the right patient.

Systemic vascular resistance is a parameter that depends on the afterload of the heart and corresponds to the resistance of the heart while it is working. It is the resistance the heart has to overcome to pump blood to the rest of the body except the lungs. The systemic vascular resistance index (SVRI) is defined as the ratio of mean arterial pressure (MAP) and central venous pressure (CVP) to cardiac index (CI) (SVRI= 80 x (MAP-CVP) / CI). In general, SVRI is proportional to MAP. It decreases due to vasodilation in septic patients. Compared to previous studies, lower SVRI in septic shock was associated with adverse outcomes and increased mortality. Invasive methods such as pulmonary artery catheters or relatively expensive methods such as PICCO are required for SVRI measurement.

Can a more cost-effective and rapid alternative to the systemic vascular resistance index measured by expensive or high-risk methods be found? Ultrasound, as modern stethoscope, is a need especially in every 3 level ICU.

The resistive index (RI) (Pourcelot index) is a noninvasive measurement used to evaluate vessel compliance with Doppler ultrasound. It is determined by a formula calculated between the systolic peak flow rate (PSV) and the end-diastolic flow rate (EDV) ((PSV-EDV)/PSV). Today RI is using for measure to assess tissue perfusion, particularly on the kidney. Renal RI shows changes in renal intravascular volume and hemodynamics. An inverse relationship has been shown between renal RI and MAP in acute kidney injury. Measurement of RI on the peripheral artery correlated with SVRI in a study of patients who had undergone cardiac surgery.

In this study the investigators will compare RI on radial artery in wrist snuffbox (SBRI) with SVRI for primary outcome. Also compare SBRI with MAP, CVP, diastolic shock index, pleth variability index, delta stroke volume index, central venous oxygen saturation (ScvO2) and partial carbon dioxide gap (Pv-aCO2) for secondary outcome.

Each patient will be followed for sepsis and septic shock. In the investigators ICU all sepsis patients has invasive artery canula for real-time monitoring and central venous catheter for blood sampling and need of vasopressor so there won't be any extra risk for this study. If a septic shock patient needs to mechanically ventilated and meets inclusion criteria, the investigators will carry out measurements just after intubation. Or, a mechanical ventilated patient who has developed septic shock; if patient has no spontaneous breathing effort, the investigators will carry out measurements. Also, arterial and central venous blood samples are taken after intubation or septic shock for every 6 hours, daily complete blood count (CBC), C-reactive protein, renal and hepatic blood analysis, and 2 times per week procalcitonin levels as routine at the hospital where the study is taking place in ICU.

Demographic parameters, physical examination notes (capillary refill time, mottling score, urine output, skin turgor), systolic, diastolic and mean arterial pressure, central venous pressure, arterial and central venous blood gas analysis, CBC and biochemistry blood analysis, Acute Physiology and Chronic Health Evaluation II (APACHE II) score, Sequential Organ Failure Assesment (SOFA) score and Nutrition Risk in the Critically Ill (NUTRIC) Score will be noted. For cardiac output monitoring Baxter Starling non-invasive monitor will be used and all hemodynamic parameters will be noted for study during examination.. For measuring SBRI Philips CX50 ultrasound device L12-3 linear probe will be used. Starling monitors 4 electrodes will be placed as specified by the manufacturer. Masimo Rad-87 probe will place hand index or middle finger. SBRI will measure for three times successive with 1.5 centimeters depth and 3 same measurement will be recorded. At the same time baseline evaluation will be started with Starling monitor and all parameters will be noted. After completion of baseline measurement Starling fluid challenge will be initiated as passive leg raising as specified by manufacturer. This procedure takes 3 minutes to calculate and after 2.5 minutes SBRI will be measured again as described above. At the end of fluid challenge all parameters will be noted.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* admitted to intensive care for septic shock
* mechanical ventilated
* non spontaneous breathing
* applied invasive artery cannulation (radial, femoral, brachial)
* applied central venous catheter (jugular, subclavian)
* SOFA score>2
* Receiving vasopressor/inotrope support to achieve MAP ≥65 mmHg
* Blood lactate >2mmol/L

Exclusion Criteria:

* <18 years old
* Hypothermia (<35C)
* Atrial fibrilation/flutter
* Pace-maker
* Severe aort valve insufficiency
* History of aortic and the great arteries adjacent to the aortic arch surgery
* Bilateral radial artery puncture in last 12 hours
* Peripheral artery disease
* Extremity amputation (leg or arm)
* Wound on forearm
* Continous Renal Replacement Therapy
* Spontaneous breath effort

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who admited to intensive care unit of Bezmialem Vakıf Univesity Hospital
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
correlation of snuffbox radial artery resistive index and systemic vascular resistance index | 1 hour. As soon as patient meets all of the inclusion criteria
  correlation of snuffbox radial artery resistive index and systemic vascular resistance index

SECONDARY OUTCOMES:
correlation of snuffbox radial artery resistive index and pleth variability index | 1 hour. As soon as patient meets all of the inclusion criteria
  correlation of snuffbox radial artery resistive index and pleth variability index
correlation of snuffbox radial artery resistive index and delta stroke volume index | 1 hour. As soon as patient meets all of the inclusion criteria
  correlation of difference in snuffbox radial artery resistive index and delta stroke volume index
correlation of snuffbox radial artery resistive index and diastolic shock index | 1 hour. As soon as patient meets all of the inclusion criteria
  correlation of snuffbox radial artery resistive index and diastolic shock index
correlation of snuffbox radial artery resistive index and central vena cava oxygen saturation and partial carbon dioxide pressure gap | 1 hour. As soon as patient meets all of the inclusion criteria
  correlation of snuffbox radial artery resistive index and central vena cava oxygen saturation and partial carbon dioxide pressure gap
correlation of snuffbox radial artery resistive index and cardiac power index | 1 hour. As soon as patient meets all of the inclusion criteria
  correlation of snuffbox radial artery resistive index and cardiac power index

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
statistical data will be shared

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Cohen J, Vincent JL, Adhikari NK, Machado FR, Angus DC, Calandra T, Jaton K, Giulieri S, Delaloye J, Opal S, Tracey K, van der Poll T, Pelfrene E. Sepsis: a roadmap for future research. Lancet Infect Dis. 2015 May;15(5):581-614. doi: 10.1016/S1473-3099(15)70112-X. Epub 2015 Apr 19. PMID 25932591
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Levy MM, Dellinger RP, Townsend SR, Linde-Zwirble WT, Marshall JC, Bion J, Schorr C, Artigas A, Ramsay G, Beale R, Parker MM, Gerlach H, Reinhart K, Silva E, Harvey M, Regan S, Angus DC. The Surviving Sepsis Campaign: results of an international guideline-based performance improvement program targeting severe sepsis. Intensive Care Med. 2010 Feb;36(2):222-31. doi: 10.1007/s00134-009-1738-3. Epub 2010 Jan 13. PMID 20069275
- [Background] Levy MM, Artigas A, Phillips GS, Rhodes A, Beale R, Osborn T, Vincent JL, Townsend S, Lemeshow S, Dellinger RP. Outcomes of the Surviving Sepsis Campaign in intensive care units in the USA and Europe: a prospective cohort study. Lancet Infect Dis. 2012 Dec;12(12):919-24. doi: 10.1016/S1473-3099(12)70239-6. Epub 2012 Oct 26. PMID 23103175
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Reuter DA, Chappell D, Perel A. The dark sides of fluid administration in the critically ill patient. Intensive Care Med. 2018 Jul;44(7):1138-1140. doi: 10.1007/s00134-017-4989-4. Epub 2017 Nov 11. No abstract available. PMID 29128963
- [Background] Kox M, Pickkers P. "Less is more" in critically ill patients: not too intensive. JAMA Intern Med. 2013 Jul 22;173(14):1369-72. doi: 10.1001/jamainternmed.2013.6702. PMID 23752755
- [Background] Groeneveld AB, Nauta JJ, Thijs LG. Peripheral vascular resistance in septic shock: its relation to outcome. Intensive Care Med. 1988;14(2):141-7. doi: 10.1007/BF00257468. PMID 3361019
- [Background] Ban K, Kochi K, Imai K, Okada K, Orihashi K, Sueda T. Novel Doppler technique to assess systemic vascular resistance: the snuffbox technique. Circ J. 2005 Jun;69(6):688-94. doi: 10.1253/circj.69.688. PMID 15914947